CLINICAL TRIAL: NCT06446869
Title: Randomised, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of the Combination of Levilactobacillus Brevis KABP-052, Lactiplantibacillus Plantarum KABP-051 and Pediococcus Acidilactici KABP-021 on Menopausal Symptoms and Quality of Life in Peri- and Post-menopausal Women
Brief Title: Menopausal Symptoms Probiotic Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Community Pharmacology Services Ltd (Other)
Collaborators: Kaneka Americas Holding Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KNK-DONACARE
Record Dates: First submitted 2024-05-17; First posted 2024-06-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Menopause
Keywords: menopause; menopausal symptoms; hot flashes; night sweats; menopause treatment
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Intervention Model Description: Study treatment vs Placebo
Who Masked: Participant, Care Provider
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gyntima Menopause (Experimental): Study treatment
  Interventions: Dietary Supplement: Gyntima Menopause
- Placebo (Placebo Comparator): Placebo comparator arm
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Gyntima Menopause — Combination of Levilactobacillus brevis KABP-052, Lactiplantibacillus plantarum KABP-051 and Pediococcus acidilactici KABP-021
  Arms: Gyntima Menopause
Other: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
In this study, we want to investigate if the active product consisting of a probiotic blend can potentiate the recirculation of active oestrogens into the bloodstream and help to mitigate menopause symptoms, which are closely related to oestrogens levels

ELIGIBILITY:
Inclusion Criteria:

* Perimenopausal or post-menopausal women with spontaneous menopause and amenorrhoea for less than 2 years
* Self reported menopausal symptoms (5 or more hot flashes/night sweats per day or 35 or more per week recorded daily for 14 consecutive days)
* BMI between 18.5 and 34.9 kg/m2
* Menopause rating score II (MRS-II) total score of 9 or more at baseline visit
* Willing to sign Informed Consent Form
* Willing to not make relevant changes to their current dietary or lifestyle habits during study
* Able to follow study procedures
* If perimenopausal, agrees to use an accepted method of contraception for duration of study.

Exclusion Criteria:

* History of hysterectomy, oophorectomy, endometrial hyperplasia, uterine or endometrial cancer, breast cancer, or cancers associated with sex hormones
* Use of hormonal replacement therapy, hormone analogues, or oral contraceptives within 3 months prior to the start of the study
* Intake of herbal or food supplements with known effects on menopause symptoms within 1 month prior to the start of the study. Examples of prohibited substances are black cohosh, melatonin, ginseng, chasteberry, phytoestrogens (e.g., hop [Humulus lupulus L.], soy isoflavones, red clover) within 1 month prior to the start of the study
* Use of any food supplement containing probiotics or postbiotics or regular consumption (>3 days/week) of foods containing probiotics (including yogurt with added probiotics or bifidus effect) within 1 month prior to the start of the study
* Use of oral (>3 days) or parenteral antibiotics within 1 month prior to the start of the study
* Participants with a new diagnosis of mental health disorder in the last 12 months or with an unstable or uncontrolled mental health disorder in the opinion of the Investigator
* Diagnosis of type 1 or uncontrolled type 2 diabetes mellitus
* Diagnosis of chronic gastrointestinal disease, such as inflammatory bowel disease (Crohn's disease or ulcerative colitis), pancreatitis, or short bowel syndrome
* History of thyroid disorders (hypothyroidism or hyperthyroidism) which are untreated or unstable
* History of gastrointestinal surgery 6 months prior to the start of the study, with the exception of appendicectomy
* Regular intake (>3 days/week) of medication that affects microbiota or bowel movements, namely laxatives like polyethylene glycol or stimulant laxatives (bisacodyl, sennosides, sodium pyrosulfate)
* History of coronary disease, myocardial infarction, unstable angina, or previous coronary angioplasty
* History of venous thromboembolism (VTE) or known to be high risk for VTE due to inherited or acquired thrombophilia (such as factor V Leiden, antiphospholipid syndrome)
* History of stroke or transient ischaemic attack
* History of severe renal dysfunction as defined by an estimated glomerular filtration rate <30 mL/minute or severe liver dysfunction defined as established cirrhosis or active liver disease with alanine aminotransferase (ALT) >3 × upper limit of normal at baseline
* Initiated for new diagnosis or changed dose of UK-approved therapeutic medication or nutraceuticals for a medical condition that can affect study outcomes according to the Investigator's judgement (i.e., statins, anti-hypertensives, etc.) within 90 days prior to study entry
* Diagnosis of primary or secondary immunodeficiency including acquired immunodeficiency syndrome, immunodeficiency, or active oncologic disease
* Known or suspected alcohol or drug abuse
* Any other surgical or medical condition, which in the opinion of the Investigator, may place the participant at higher risk from her participation in the study, or is likely to prevent the participant from complying with the requirements of the study or completing the study
* Currently participating in another study or having participated in one within 3 months prior to the start of the study
* The participant is pregnant, planning a pregnancy, or breastfeeding

Ages: 42 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-07-25 (Estimated); Study Completion 2026-10-25 (Estimated)

PRIMARY OUTCOMES:
Assess Impact | 120 days
  To assess the impact of the investigational product on the symptoms and quality of life (QoL) in menopausal women as assessed by Menopause Rating Score II (MRS-II) Each of the 11 symptoms contained in the scale can get 0 (no complaints) or up to 4 scoring points (severe symptoms) depending on the severity of the complaints perceived by the women completing the scale (an appropriate box is to be ticked). The score increases point by point with increasing severity of subjectively perceived symptoms in each of the 11 items.

SECONDARY OUTCOMES:
Impact on Severity of Symptoms | 120 days
  To assess the impact of the investigational product on the severity of symptoms as assessed by MRS-II
  Each of the 11 symptoms contained in the scale can get 0 (no complaints) or up to 4 scoring points (severe symptoms) depending on the severity of the complaints perceived by the women completing the scale (an appropriate box is to be ticked). The score increases point by point with increasing severity of subjectively perceived symptoms in each of the 11 items.
Impact on number of Hot Flashes / Night Sweats | 120 days
  To assess the impact of the investigational product on the number of hot flashes and night sweats.
  All study participants will receive a diary where they will report their daily number of hot flashes and night sweats.
Impact on Intensity of Hot Flashes / Night Sweats | 120 days
  To assess the impact of the investigational product on the intensity of hot flashes and night sweats
  All study participants will receive a diary where they will report their daily number of hot flashes and night sweats.
Impact on QoL | 120 days
  To assess the impact of the investigational product on menopause-related QoL as assessed by the Greene Climacteric Scale (GCS) questionnaire
  The Greene Climacteric Scale (GCS) is a standard list of 21 questions which women use to rate how much they are bothered by menopause symptoms such as hot flashes, night sweats, rapid heartbeat, and difficulty sleeping. Each symptom is rated on a 4-point Likert scale from 0 points (not at all) to 3 points (Extremely)
Impact on Depression, Anxiety and Stress | 120 days
  To assess the impact of the investigational product on Depress, Anxiety and Stress Scale-21 (DASS-21)
  This scale form is a short form of the 42 item self reported questionnaire measuring depression, anxiety and stress. The 21 items on this questionnaire comprise a set of 3 self-reported scales designed to assess DASS. The 7 elements on the scales are graded on a Likert scale from 0 to 3.
Impact on levels of reproductive hormones | 120 days
  To assess the impact of the investigational product on levels of relevant reproductive hormones during peri- and post-menopause
  Efficacy laboratory tests are to be performed for all participants as indicated in the protocol's SoA. For Hormones - Oestrone, Oestradiol, FSH and progesterone.
Impact on serum inflammation markers | 120 days
  To assess the impact of the investigational product on serum inflammation markers
  Efficacy laboratory tests are to be performed for all participants, as indicated in the protocol's SoA. For Biomarkers - Interleukin (IL)-1β, IL-2, IL-4, IL-6, IL-8, tumour necrosis factor (TNF) and interferon). Note: Analysis of inflammation biomarkers will only be performed at the Sponsor's discretion after the results of hot flashes and QoL become available.
Impact on gut microbiota composition | 120 days
  To assess the impact of the investigational product on gut microbiota composition
  The determination of the composition of the faecal microbiota will be carried out through a study of the V3-V4 hypervariable regions of the bacterial ribosomal 16S rRNA gene. Next, the libraries will be set up, and ultrasequencing, bioinformatics and statistical analysis will be carried out. The analysis will be performed in a specialised company called Microomics Systems S.L. located in Barcelona, Spain. Stool samples will be collected by study participants
Impact on digestive tolerance | 120 days
  To assess the impact of the investigational product on digestive tolerance.
  This will be assessedbased on documented gastrointestinal symptoms on the Gastrointestinal Symptom Rating Scale (GSRS)
Safety of the IP | 120 days
  To assess the safety of the investigational product Safety evaluation based on AE registry, Blood cell count and basic blood biochemistry
Satisfaction of Use | 120 days
  To assess the satisfaction with the use of the investigational product
  Product satisfaction will be evaluated by using an ordinal 5-point Likert scale, where study participants will have to rate the degree to which they agree or disagree with the statement: "Please indicate the degree of satisfaction or dissatisfaction with the way the study product has relieved your symptoms associated to menopause"

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Laing, MBChB, Principal Investigator — Community Pharmacology Services Ltd
Locations (1):
- FutureMeds Glasgow, Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No data will be shared